CLINICAL TRIAL: NCT01392521
Title: Phase Ib Trial of the Combination of PI3K Inhibitor BAY 80-6946 and Allosteric-MEK Inhibitor BAY 86-9766 in Subjects With Advanced Cancer
Brief Title: Phase Ib Study of PI3(Phosphoinositol 3)-Kinase Inhibitor Copanlisib With MEK (Mitogen-activated Protein Kinase) Inhibitor Refametinib (BAY86-9766) in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12876; 2010-024082-45 (EudraCT Number)
Record Dates: First submitted 2011-06-30; First posted 2011-07-12 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Neoplasms
Keywords: Safety; Tolerability; Pharmacokinetics
MeSH Terms: conditions — Neoplasms | interventions — copanlisib; N-(3,4-difluoro-2-(2-fluoro-4-iodophenylamino)-6-methoxyphenyl)-1-(2,3-dihydroxypropyl)cyclopropane-1-sulfonamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Copanlisib + Refametinib (BAY86-9766)

INTERVENTIONS:
Drug: Copanlisib + Refametinib (BAY86-9766) — Copanlisib will be administered as an IV infusion weekly for 3 weeks in combination with Refametinib (BAY86-9766) at varying dose levels. Refametinib (BAY86-9766) is administered orally twice a day starting at Day 4 of Cycle 1.
Drug: Copanlisib + Refametinib (BAY86-9766) — Copanlisib will be administered as an IV infusion weekly in combination with Refametinib (BAY86-9766) at varying dose levels. Refametinib (BAY86-9766) is administered orally twice a day starting at Day 6 of Cycle 1 on a 4 day on, 3 day off schedule.

SUMMARY:
The PI3K (phosphoinositol 3-Kinase) inhibitor Copanlisib and the MEK (mitogen-activated protein kinase) inhibitor Refametinib (BAY86-9766)have both been tested as single agent treatments in other phase I studies. This study will test the combination of these two drugs to try and answer the following questions:

1. What are the side effects of the combination of Copanlisib and Refametinib (BAY86-9766)when given together at different/increasing dose levels?
2. What dose level of Copanlisib and Refametinib (BAY86-9766) should be tested in future clinical research studies?
3. How much Copanlisib is in the blood at specific times after administration and does adding Refametinib (BAY86-9766) have an affect?
4. How much Refametinib (BAY86-9766) is in the blood at specific times after administration and does adding Copanlisib have an affect?
5. Does the combination of Refametinib (BAY86-9766) and Copanlisib have an effect on tumors?

ELIGIBILITY:
Inclusion Criteria:

* Age greater than/equal to 18 years old
* ECOG Performance Status of 0 - 1
* Life expectancy of at least 12 weeks
* Patients with advanced, histologically or cytologically confirmed solid tumors, refractory to any standard therapy or have no standard therapy available
* LVEF (left ventricular ejection fraction) > or = to the lower limit of normal for the institution
* Radiographically or clinically evaluable tumor
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 14 days prior to start of first dose:

  * Hemoglobin > 9.0 g/dL
  * Absolute neutrophil count (ANC) > or = 1500/mm3
  * Platelet count > or = 100,000 /mm3
  * Total bilirubin < or = 1.5 times the upper limit of normal
  * ALT (alanine aminotransferase) and AST (aspartate aminotransferase) < or = 2.5 x upper limit of normal (< or = 5 x upper limit of normal for patients with liver involvement)
  * PT-INR (prothrombin-international normalized ratio) and PTT (partial thromboplastin time) < or = 1.5 times the upper limit of normal
  * Serum creatinine < or = 1.5 times the upper limit of normal

Exclusion Criteria:

* History of impaired cardiac function or clinically significant cardiac disease (i.e. congestive heart failure (CHF) NYHA (New York Heart Association) Class III or IV); active coronary artery disease, myocardial infarction within 6 months of study entry; new onset or unstable angina within 3 months of study entry, or cardiac arrhythmias requiring anti-arrhythmic therapy
* Type 1 or type 2 diabetes mellitus or fasting glucose > 125 mg/dL or HgBA1c > or = 7.0
* Use of systemic corticosteroids within 2 weeks of study entry
* History of retinal vein occlusion
* Known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Active clinically serious infection
* Uncontrolled hypertension
* Positive for HIV, or chronic Hepatitis B or C
* Subjects undergoing renal dialysis
* Known bleeding diathesis
* Ongoing substance abuse
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-07; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 2 years
Comparison of the Copanlisib AUC when given alone with the AUC when given with Refametinib (BAY86-9766) | At day 15
Comparison of the Refametinib (BAY86-9766) AUC when given alone with the AUC when given with Copanlisib | At day 15

SECONDARY OUTCOMES:
Tumor Response as measured by RECIST 1.1 criteria | 3 years
Biomarker evaluation including analysis of pathway activation in blood and plasma | 3 years
Tumor Response as measured by FDG-PET at MTD and expansion cohort(s) | 3 years
Pharmacodynamic biomarker evaluation analysis using paired tumor biopsies | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (8):
- United States (6):
  - Scottsdale, Arizona
  - Las Vegas, Nevada
  - Greenville, South Carolina
  - Houston, Texas
  - Tyler, Texas
  - Vancouver, Washington
- Freiburg im Breisgau, Baden-Wurttemberg, Germany
- Rotterdam, Netherlands

REFERENCES:
- [Derived] Ramanathan RK, Von Hoff DD, Eskens F, Blumenschein G Jr, Richards D, Genvresse I, Reschke S, Granvil C, Skubala A, Pena C, Mross K. Phase Ib Trial of the PI3K Inhibitor Copanlisib Combined with the Allosteric MEK Inhibitor Refametinib in Patients with Advanced Cancer. Target Oncol. 2020 Apr;15(2):163-174. doi: 10.1007/s11523-020-00714-0. PMID 32314268